CLINICAL TRIAL: NCT03936166
Title: A Double-Blind, Randomized, Placebo-Controlled, Single- And-Multiple-Ascending Dose Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of CRN01941 in Healthy Volunteers
Brief Title: A Single and Multiple-Ascending Dose Study of CRN01941 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Crinetics Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRN01941-01
Record Dates: First submitted 2019-04-25; First posted 2019-05-03 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: Single and multiple-dose cohorts are placebo-controlled.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single Ascending Dose (Part 1) (Experimental)
  Interventions: Drug: CRN01941 Oral Solution; Drug: CRN01941 Oral Capsule; Drug: Placebo Oral Solution; Drug: Placebo Oral Capsule
- Multiple Ascending Dose (Part 2) (Experimental)
  Interventions: Drug: CRN01941 Oral Solution; Drug: CRN01941 Oral Capsule; Drug: Placebo Oral Solution; Drug: Placebo Oral Capsule
- Elderly Cohort (Part 3) (Placebo Comparator)
  Interventions: Drug: CRN01941 Oral Solution; Drug: CRN01941 Oral Capsule; Drug: Placebo Oral Solution; Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: CRN01941 Oral Solution — Investigational drug
Drug: CRN01941 Oral Capsule — Investigational drug
Drug: Placebo Oral Solution — Placebo
Drug: Placebo Oral Capsule — Placebo

SUMMARY:
This is a Phase 1, double-blind, randomized, placebo-controlled, single-dose and multiple-dose study of CRN01941 in up to 119 healthy male and female subjects. This single-center study will be conducted in 3 parts: a single-ascending dose phase (up to 8 cohorts, 8 subjects/cohort), a multiple-ascending dose phase (up to 5 cohorts, 9 subjects/cohort), and single dose phase in elderly subjects (1 cohort, 10 subjects).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects 18 to 55 years of age, inclusive, at time of screening (Parts 1 and 2 only).
2. Males and females subjects 65 to 85 years of age at screening (Part 3 only).
3. Females must be non-pregnant and non-lactating, postmenopausal by history and confirmed by follicle stimulating hormone (FSH) >30 U/L at Screening, or surgically sterile.
4. Male subjects must be surgically sterile or agree to use highly effective form of contraception when sexually active with a female partner of child bearing potential.
5. Body mass index (BMI) of 18 to 32 kg/m2, inclusive at Screening.
6. Willing to provide signed informed consent.

Exclusion Criteria:

1. Any uncontrolled or active major systemic disease which makes study participation unsafe or could interfere with evaluation of the endpoints of the study.
2. History or presence of malignancy within the past 5 years, not including treated basal cell carcinomas and in situ cervical neoplasia.
3. Use of any investigational drug within the past 60 days.
4. Have a medically significant abnormality observed during screening or admission.
5. Use of any prior medication without approval of the investigator within 14 days prior to admission.
6. Subjects with human immunodeficiency virus (HIV), hepatitis B or hepatitis C infections. Subjects with previous hepatitis C infection that is now cured may be eligible.
7. History of or current alcohol or substance abuse in the past 12 months
8. Any condition that in the opinion of the investigator would jeopardize the subject's appropriate participation in this Phase 1 study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events by severity | Part 1 - up to Day 8; Part 2 - up to Day 20; Part 3 - up to Day 8
Number of participants with serious adverse events (SAEs) | Part 1 - up to Day 8; Part 2 - up to Day 20; Part 3 - up to Day 8
Number of participants with clinically significant changes in vital signs | Part 1 - up to Day 8; Part 2 - up to Day 20; Part 3 - up to Day 8
Number of participants with ECG abnormalities | Part 1 - up to Day 8; Part 2 - up to Day 20; Part 3 - up to Day 8
Number of participants with clinical laboratory abnormalities | Part 1 - up to Day 8; Part 2 - up to Day 20; Part 3 - up to Day 8

SECONDARY OUTCOMES:
Pharmacokinetics (AUC) | Part 1 - up to Day 8; Part 2 - up to Day 20; Part 3 - up to Day 8
  Assessment of the plasma area under the curve of CRN01941
Pharmacokinetics (Cmax) | Part 1 - up to Day 8; Part 2 - up to Day 20; Part 3 - up to Day 8
  Assessment of the maximum observed plasma concentration of CRN01941
Pharmacokinetics (Tmax) | Part 1 - up to Day 8; Part 2 - up to Day 20; Part 3 - up to Day 8
  Assessment of the time to reach Cmax for CRN01941
Pharmacokinetics (T1/2) | Part 1 - up to Day 8; Part 2 - up to Day 20; Part 3 - up to Day 8
  Assessment of the elimination half-life of CRN01941

CONTACTS AND LOCATIONS:
Locations (1):
- Linear Clinical Research, Perth, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No